CLINICAL TRIAL: NCT02906709
Title: A Phase IV, Multicenter, Randomized, Placebo-Controlled, Parallel-Group, Double-Blind Trial and Subsequent Open-Label, Extension Trial to Assess the Safety and Efficacy of Addition of Omarigliptin in Japanese Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Insulin Monotherapy in Addition to Diet and Exercise Therapy
Brief Title: Omarigliptin Add-on to Insulin in Japanese Participants With Type 2 Diabetes Mellitus (T2DM, MK-3102-039)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3102-039; MK-3102-039 (Other: Merck Protocol Number); 163455 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omarigliptin 25 mg (Experimental): Omarigliptin 25 mg once weekly for 52 weeks (Phase A and B)
  Interventions: Drug: Omarigliptin; Biological: Insulin
- Placebo→Omarigliptin 25 mg (Experimental): Placebo to Omarigliptin once weekly for 16 weeks (Phase A) switching to Omarigliptin 25 mg once weekly for 36 weeks (Phase B)
  Interventions: Drug: Omarigliptin; Drug: Placebo; Biological: Insulin

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin, 25 mg orally once weekly
  Other Names: MK-3102; MARIZEV®
Drug: Placebo — Placebo to omarigliptin orally once weekly
  Arms: Placebo→Omarigliptin 25 mg
Biological: Insulin — Insulin will be administered subcutaneously during the trial as monotherapy; dosage and administration following each package insert.

SUMMARY:
This study will examine the efficacy of omarigliptin 25 mg once weekly compared to placebo in Japanese patients with T2DM who have inadequate glycemic control on insulin monotherapy in addition to diet and exercise therapy. The primary hypothesis of the study is that omarigliptin 25 mg once weekly provides greater reduction in hemoglobin A1C (HbA1c) compared with placebo as assessed by change from baseline to Week 16 [Phase A (double-blind period)].

DETAILED DESCRIPTION:
After a screening period of up to 2 weeks followed by a pretreatment period of 2 or 10 weeks, each participant will be receiving assigned double-blind treatment (omarigliptin 25 mg or placebo once weekly) for approximately 16 weeks (Phase A) followed by 36 weeks of open-label treatment (omarigliptin 25 mg once weekly, Phase B). After the end of treatment each participant will be followed for 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM
* Meet all of following criteria at Week -2 of pre-randomization

  1. On diet and exercise therapy for 6 weeks or longer, AND
  2. Have been on a stable dosage and administration of insulin (8 to 40 units/day) for 10 weeks or longer, AND.
  3. Have not been on any additional anti-hyperglycemic agent (AHAs, except for insulin monotherapy) for 8 weeks or longer, AND
  4. HbA1c ≥7.5% and ≤10.0%
  5. Fasting Plasma Glucose (FPG) ≥126 mg/dL and ≤230 mg/dL
* Have a body mass index (BMI) >18 kg/m^2 and <40 kg/m^2
* A male or female not of reproductive potential or a female of reproductive potential and agrees to remain abstinent from heterosexual activity, or agrees to use acceptable contraception to prevent pregnancy.

Exclusion Criteria:

* Has type 1 diabetes mellitus or has a history of diabetic ketoacidosis.
* Has a history of being administered any of the following AHAs including fixed dose combination (FDC) containing the following ingredients:

  1. Thiazolidinediones within 12 weeks
  2. Glucagon-like peptide 1 (GLP-1) receptor agonists within 12 weeks
  3. Omarigliptin at any time
* Has history of severe hypoglycemia with coma or loss of consciousness, or for whom hypoglycemia was observed greater or equal to two times per week within 8 weeks
* Is currently participating in or has participated in another study with an investigational compound or device within the prior 12 weeks
* Has undergone a surgical procedure within 8 weeks or has planned major surgery during the study.
* Receives a lipid-lowering medication or thyroid replacement therapy at unstable dosage and administration
* Has poorly controlled hypertension
* Has a medical history of active liver disease, including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease.
* Has human immunodeficiency virus (HIV).
* Has had new or worsening signs or symptoms of coronary heart disease or congestive heart failure within the past 3 months, or has acute coronary syndrome, coronary artery intervention, or stroke or transient ischemic neurological disorder within the past 3 months
* Has severe peripheral vascular disease.
* Has a history of malignancy ≤ 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer:
* Has a clinically important hematological disorder.
* (For women of childbearing potential) has a positive urine pregnancy test.
* Is pregnant or breast feeding
* Is expected to conceive during the study
* Is expected to undergo hormonal therapy in preparation to donate eggs during the study
* Routinely consumes >14 alcoholic drinks per week or engages in binge drinking
* Has donated or plans to donate blood products of >300 mL within 8 weeks or during the study
* Has received or plans to receive blood products within 12 weeks or during the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Kadowaki T, Seino Y, Kaku K, Okamoto T, Kameya M, Sato A, Hirano T, Oshima N, Gantz I, O'Neill EA, Engel SS; Omarigliptin Study 039 Group. A randomized, placebo-controlled study to evaluate the efficacy and safety of adding omarigliptin to insulin therapy in Japanese patients with type 2 diabetes and inadequate glycaemic control. Diabetes Obes Metab. 2021 Jun;23(6):1242-1251. doi: 10.1111/dom.14331. Epub 2021 Feb 17. PMID 33512755

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo→Omarigliptin 25 mg: Placebo once weekly for 16 weeks (Phase A) switching to Omarigliptin 25 mg once weekly for 36 weeks (Phase B)
Period: Phase A (Week 0 to Week 16)
Arm/Group | Omarigliptin 25 mg | Placebo→Omarigliptin 25 mg
Started | 123 | 61
Completed | 122 | 58
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Death | 0 | 1
Period: Phase B (Extension, Week 17 to Week 52)
Arm/Group | Omarigliptin 25 mg | Placebo→Omarigliptin 25 mg
Started | 122 | 58
Completed | 117 | 58
Not Completed | 5 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omarigliptin 25 mg | Placebo→Omarigliptin 25 mg | Total
Number analyzed (Participants) | 123 | 61 | 184
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (11.0) | 60.9 (11.7) | 61.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 14 | 51
  Male | 86 | 47 | 133
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 123 | 61 | 184
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Hemoglobin A1C [Mean (Standard Deviation); unit: Percent A1C] — Hemoglobin A1C (A1C) is a measure of the percentage of glycated hemoglobin in the blood. Baseline values of A1C are presented.
  Percent A1C | 8.81 (0.68) | 8.83 (0.78) | 8.82 (0.71)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Blood glucose was measured on a fasting basis. Baseline values of FPG are expressed as mg/dL.
  mg/dL | 159.1 (31.9) | 152.2 (26.0) | 156.8 (30.2)
Baseline 1,5-anhydroglucitol (1,5-AG) Levels [Mean (Standard Deviation); unit: mg/L] — 1,5-anhydroglucitol (1,5-AG) is a marker of short-term glycemic control especially postprandial hyperglycemia. Baseline values of 1,5-AG are presented.
  mg/L | 3.6 (2.7) | 3.4 (2.1) | 3.5 (2.5)
Prior Antihyperglycemic Therapy Status [Count of Participants; unit: Participants] — The number of participants receiving antihyperglycemic therapy at baseline are presented.
  Participants
    Yes | 43 | 22 | 65
    No | 80 | 39 | 119

OUTCOME MEASURES:

1. Primary Outcome: Constrained Longitudinal Data Analysis of Change From Baseline in Hemoglobin A1c (HbA1c) at Week 16 Excluding Data After Glycemic Rescue (Phase A)
Description: HbA1c is a measure of the percentage of glycated hemoglobin in the blood. Participant whole blood samples were collected at baseline and Week 16 to determine the Constrained Longitudinal Data Analysis least squares mean HbA1c change from baseline (i.e., HbA1c at Week 16 minus HbA1c at baseline). Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. Data after glycemic rescue were excluded from this analysis. Negative data values indicated a reduction in HbA1c levels.
Time Frame: Baseline (Day 1) and Week 16
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment and had at least one measurement (baseline or post randomization) for the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent HbA1c
Groups:
- Omarigliptin 25 mg: Omarigliptin 25 mg once weekly for 16 weeks (Phase A)
- Placebo: Placebo once weekly for 16 weeks (Phase A)
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 123 | 61
Percent HbA1c | -0.61 [-0.75 to -0.47] | 0.29 [0.09 to 0.49]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -0.90, 95% CI 2-sided [-1.15 to -0.66]; Based on a Constrained Longitudinal Data Analysis model with terms for treatment, prior AHA therapy status (yes/no), time and the interaction of time by treatment, time by prior anti-hyperglycemic agent (AHA) therapy status and time by treatment by prior AHA status with the restriction of a common baseline mean between two treatment groups

2. Primary Outcome: Percentage of Participants Who Experienced One or More Adverse Events (AE) Excluding Data After Glycemic Rescue (Phase A)
Description: An adverse event is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. Data after glycemic rescue were excluded from this analysis.
Time Frame: Up to Week 16
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment and had safety data for the specified measurement and timeframe.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 123 | 61
Percentage of participants | 51.2 | 44.3
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority; Difference in % vs. Placebo = 7.0, 95% CI 2-sided [-8.4 to 21.8]; Based on Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants Who Experienced One or More AE (Omarigliptin [Phase A+B]; Placebo→Omarigliptin [Phase B Only])
Description: An adverse event is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. The results for the Placebo→Omarigliptin group summarized data from the open label period only (36 weeks), which corresponds to the study interval in which those participants were exposed to omarigliptin.
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Groups:
- Omarigliptin 25 mg (Phase A and B): Omarigliptin 25 mg once weekly for 52 weeks (Phase A and B)
- Placebo→Omarigliptin 25 mg (Phase B Only): Omarigliptin 25 mg once weekly for 36 weeks (Phase B, Week 17 to Week 52) after switching from placebo
Arm/Group | Omarigliptin 25 mg (Phase A and B) | Placebo→Omarigliptin 25 mg (Phase B Only)
Number analyzed (Participants) | 123 | 58
Percentage of Participants | 84.6 | 67.2

4. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE Excluding Data After Glycemic Rescue (Phase A)
Description: as for outcome 2
Time Frame: Up to Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 123 | 61
Percentage of Participants | 0.8 | 4.9
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority; Difference in % vs. Placebo = -4.1, 95% CI 2-sided [-12.8 to 0.4]; Based on Miettinen & Nurminen method

5. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE Including Data After Glycemic Rescue (Omarigliptin [Phase A+B]; Placebo→Omarigliptin [Phase B Only])
Description: as for outcome 3
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Omarigliptin 25 mg (Phase A and B) | Placebo→Omarigliptin 25 mg (Phase B Only)
Number analyzed (Participants) | 123 | 58
Percentage of Participants | 3.3 | 0

6. Secondary Outcome: Constrained Longitudinal Data Analysis of Change From Baseline in Fasting Plasma Glucose (FPG) at Week 16 Excluding Data After Glycemic Rescue (Phase A)
Description: Blood glucose was measured on a fasting basis. FPG is expressed as mg/dL. Blood was drawn at predose on Day 1 and after 16 weeks of treatment to determine Constrained Longitudinal Data Analysis change in plasma glucose levels (i.e., FPG at Week 16 minus FPG at baseline). Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. Data after glycemic rescue were excluded from this analysis. Negative data values indicated a reduction in FPG levels.
Time Frame: Baseline (Day 1) and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 123 | 61
mg/dL | -11.6 [-17.5 to -5.7] | 3.4 [-4.7 to 11.5]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority; p = 0.002, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -15.0, 95% CI 2-sided [-24.5 to -5.4]; Based on a Constrained Longitudinal Data Analysis model with terms for treatment, prior AHA therapy status (yes/no), time and the interaction of time by treatment, time by prior AHA therapy status and time by treatment by prior AHA status with the restriction of a common baseline mean between two treatment groups

7. Secondary Outcome: Percentage of Participants Achieving Hemoglobin A1c Goals (<7.0%) at Week 16 Constrained Longitudinal Data Analysis Using Multiple Imputation Excluding Data After Glycemic Rescue (Phase A)
Description: HbA1c is a measure of the percentage of glycated hemoglobin in the blood. Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. Data after glycemic rescue were excluded from this analysis. Each of the 10 imputed data sets was summarized to obtain the percentage of responders within each group and were combined using standard multiple imputation techniques to yield an overall estimate of response rate and associated variance for each group. A constrained longitudinal data analysis was used to analyze the data and Wilson score method by treatment groups used for the analysis of percentages of individuals at the HbA1c goals of <7.0% at Week 16 and the 95% confidence intervals (CIs). Miettinen & Nurminen (M&N) method after imputations were used to calculate the treatment differences of the percentages of individuals and the 95% CIs.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 123 | 61
Percentage of Participants | 5.8 [2.8 to 11.5] | 0.0 [0.0 to 6.2]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority; p = 0.065, Miettinen & Nurminen method; Percent Between-group Rate Difference = 5.8, 95% CI 2-sided [-0.7 to 11.5]; The estimated response rates and effective sample sizes were used to obtain the confidence intervals (CIs) for within-group response rates via the Wilson score method. The CI were calculated via the stratified (non-combination prior AHA therapy status) Miettinen & Nurminen method

8. Secondary Outcome: Percentage of Participants Achieving HbA1c Goals (<6.5%) at Week 16 Constrained Longitudinal Data Analysis Using Multiple Imputation Excluding Data After Glycemic Rescue (Phase A)
Description: HbA1c is a measure of the percentage of glycated hemoglobin in the blood. Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. Data after glycemic rescue were excluded from this analysis. Each of the 10 imputed data sets was summarized to obtain the percentage of responders within each group and were combined using standard multiple imputation techniques to yield an overall estimate of response rate and associated variance for each group. A constrained longitudinal data analysis was used to analyze the data and Wilson score method by treatment groups used for the analysis of percentages of individuals at the HbA1c goals of <6.5% at Week 16 and the 95% confidence intervals (CIs). Miettinen & Nurminen (M&N) method after imputations were used to calculate the treatment differences of the percentages of individuals and the 95% CIs.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 123 | 61
Percentage of Participants | 1.7 [0.4 to 5.9] | 0.0 [0.0 to 6.2]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority; p = 0.334, Miettinen & Nurminen method; Percent Between-group Rate Difference = 1.6, 95% CI 2-sided [-4.7 to 5.8]; [other analysis details as in outcome 7, analysis 1]

9. Secondary Outcome: Constrained Longitudinal Data Analysis of Change From Baseline in 1,5-anhydroglucitol (1,5-AG) at Week 16 Excluding Data After Glycemic Rescue (Phase A)
Description: 1,5-anhydroglucitol (1,5-AG) is a marker of short-term glycemic control especially postprandial hyperglycemia. 1,5-AG accurately predicts rapid changes in glycemia and is tightly associated with glucose fluctuations and postprandial glucose. Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. Data after glycemic rescue were excluded from this analysis. Data (1,5-AG at Week 16 minus 1,5-AG at baseline) was analyzed by Constrained Longitudinal Data Analysis. Positive data values indicate an increase in 1,5-AG levels and correlate with an improvement in glycemia.
Time Frame: Baseline (Day 1) and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 123 | 61
mg/L | 2.9 [2.4 to 3.4] | -0.2 [-0.9 to 0.5]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = 3.1, 95% CI 2-sided [2.3 to 4.0]; [other analysis details as in outcome 6, analysis 1]

10. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 52 (Phase A+B)
Description: HbA1c is a measure of the percentage of glycated hemoglobin in the blood. Participant whole blood samples were collected at baseline and Week 52 to determine the mean HbA1c change from baseline (i.e., HbA1c at Week 52 minus HbA1c at baseline). Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. Negative data values indicated a reduction in HbA1c levels.
Time Frame: Baseline (Day 1) and Week 52
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment and had at least one measurement (baseline or post randomization) for the outcome measure. Three participants in the Placebo group did not have data to contribute to the analysis.
Measure: Mean (95% Confidence Interval); unit: Percent A1C
Arm/Group | Omarigliptin 25 mg | Placebo→Omarigliptin 25 mg
Number analyzed (Participants) | 123 | 58
Percent A1C | -0.57 [-0.73 to -0.42] | -0.57 [-0.81 to -0.32]

11. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52 (Phase A+B)
Description: Blood glucose was measured on a fasting basis. FPG is expressed as mg/dL. Blood was drawn at predose on Day 1 and after 52 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 52 minus FPG at baseline). Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. Negative data values indicated a reduction in FPG levels.
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 25 mg | Placebo→Omarigliptin 25 mg
Number analyzed (Participants) | 123 | 58
mg/dL | -11.5 [-18.6 to -4.5] | -5.3 [-14.1 to 3.6]

12. Secondary Outcome: Percentage of Participants Achieving Hemoglobin A1c Goals (<7.0%) at Week 52 (Phase A+B)
Description: HbA1c is a measure of the percentage of glycated hemoglobin in the blood. Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. For the HbA1c goals of <7.0% at Week 52, the percentage of participants and the 95% confidence intervals were calculated using Wilson score method by treatment groups of the double-blind period.
Time Frame: Week 52
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment and had at least one measurement (baseline or post randomization). Three participants in the Placebo group did not have data to contribute to the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Omarigliptin 25 mg | Placebo→Omarigliptin 25 mg
Number analyzed (Participants) | 123 | 58
Percentage of Participants | 7.3 [3.9 to 13.3] | 8.6 [3.7 to 18.6]

13. Secondary Outcome: Percentage of Participants Achieving Hemoglobin A1c Goals (<6.5%) at Week 52 (Phase A+B)
Description: HbA1c is a measure of the percentage of glycated hemoglobin in the blood. Participants that met rescue criteria had their insulin dose adjusted as determined clinically appropriate by the investigator to manage glycemic control. For the HbA1c goals of <6.5% at Week 52, the percentage of participants and the 95% confidence intervals were calculated using Wilson score method by treatment groups of the double-blind period.
Time Frame: Week 52
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Omarigliptin 25 mg | Placebo→Omarigliptin 25 mg
Number analyzed (Participants) | 123 | 58
Percentage of Participants | 1.6 [0.4 to 5.7] | 0.0 [NA to NA] — Since no participants achieved a HbA1c goal of <6.5% at Week 52, no confidence intervals could be calculated.

ADVERSE EVENTS:
Time Frame: Phase A (Up to 16 weeks), Phase B (Up to 36 weeks [Week 17 to 52]), Phase A+B (Up to 52 weeks)
Description: The analysis population consisted of all randomized participants who received at least one dose of study treatment and had safety data for the specified timeframe. Adverse Events include data after glycemic rescue. The results for the Placebo→Omarigliptin (Phase B only) group summarize data from the open-label period only (36 weeks), which corresponds to the study interval in which participants were exposed to omarigliptin.
Groups:
- Omarigliptin 25 mg (Phase A): Omarigliptin 25 mg once weekly for 16 weeks (Phase A)
- Placebo (Phase A): Placebo once weekly for 16 weeks (Phase A)
- Omarigliptin 25 mg (Phase A + B): Omarigliptin 25 mg once weekly for 52 weeks (Phase A and B)
- Placebo→Omarigliptin (Phase B Only): Omarigliptin 25 mg once weekly for 36 weeks (Phase B) after switching from placebo
Arm/Group | Omarigliptin 25 mg (Phase A) | Placebo (Phase A) | Omarigliptin 25 mg (Phase A + B) | Placebo→Omarigliptin (Phase B Only)
All-Cause Mortality (participants affected / at risk) | 0/123 | 1/61 | 0/123 | 0/58
Serious Adverse Events (participants affected / at risk) | 5/123 | 2/61 | 12/123 | 1/58
Other Adverse Events (participants affected / at risk) | 35/123 | 11/61 | 72/123 | 27/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 25 mg (Phase A) (N=123) | Placebo (Phase A) (N=61) | Omarigliptin 25 mg (Phase A + B) (N=123) | Placebo→Omarigliptin (Phase B Only) (N=58)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 25 mg (Phase A) (N=123) | Placebo (Phase A) (N=61) | Omarigliptin 25 mg (Phase A + B) (N=123) | Placebo→Omarigliptin (Phase B Only) (N=58)
Nasopharyngitis (Infections and infestations) | 12 (13) | 5 (5) | 40 (60) | 20 (28)
Hypoglycaemia (Metabolism and nutrition disorders) | 18 (28) | 5 (11) | 30 (98) | 8 (17)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 8 (10) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 0 (0) | 7 (8) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 7 (8) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 8 (10) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT02906709/Prot_SAP_000.pdf